CLINICAL TRIAL: NCT00006326
Title: A Randomized, Open-Label Study to Evaluate 3 Salvage Regimens in HIV-Infected Subjects Experiencing Virologic Failure on an Initial HAART Regimen Containing Nelfinavir
Brief Title: Safety and Effectiveness of 3 Anti-HIV Treatments in Patients Who Have Failed Previous Treatments Containing Nelfinavir
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 228H; AG1343-1133; 1133
Record Dates: First submitted 2000-10-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Delavirdine; Reverse Transcriptase Inhibitors; Salvage Therapy; Anti-HIV Agents; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Delavirdine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Delavirdine mesylate

SUMMARY:
The purpose of this study is to see if 3 anti-HIV drug combinations are safe and effective in patients who have failed previous anti-HIV treatments using nelfinavir (NFV).

DETAILED DESCRIPTION:
Patients receive 1 of 3 salvage regimens. Treatments A and B include delavirdine, 1 of 2 doses of indinavir, and 2 nucleoside reverse transcriptase inhibitors (NRTIs) to which the patient has not been exposed. Treatment C includes ritonavir, indinavir, and 2 NRTIs to which the patient has not been exposed. When virologic failure is first observed, the patient must return in 2 weeks for confirmation of failure and start the salvage regimen within 1 month of the first assay in which failure was observed. Patients who have less than 400 copies/ml HIV RNA after 16 weeks of therapy are considered responders and continue on the study. Those who have more than 400 copies/ml after 16 weeks of therapy are considered nonresponders and should be discontinued from the study. In addition, patients who respond and subsequently rebound with a viral load 0.5 log above the nadir and greater than 400 copies/ml on 2 consecutive assays at least 2 weeks apart are considered treatment failures and should be discontinued from the study. Patients have regular physical exams, as well as virologic, immunologic, and pharmacokinetic assessments.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Had a viral load of less than 400 copies/ml, followed by an increase in viral load while taking an anti-HIV drug combination including NFV (treatment failure).
* Can start the study treatment within 1 month of treatment failure.
* Have a viral load of less than 30,000 copies/ml when they enter the study.
* Have not taken nonnucleoside reverse transcriptase inhibitors (NNRTIs) or protease inhibitors (PIs) other than NFV.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- Susan Conner, San Diego, California, United States